CLINICAL TRIAL: NCT00540813
Title: Paclitaxel-Eluting Balloon Angioplasty and Coroflex™-Stents in the Treatment of Bifurcated Coronary Lesions
Acronym: PEPCAD V
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heart Centre Rotenburg (Other)
Collaborators: B. Braun Melsungen AG (Industry); Clinical Research Institute Rotenburg a.d.F. (Unknown)
Responsible Party: Principal Investigator, Ralf Degenhardt, PhD, Data Manager, Heart Centre Rotenburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBM-VS-56
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Ischemia; Stenosis
Keywords: bifurcation stenosis; Patients with documented ischemia due to a de-novo bifurcation stenosis
MeSH Terms: conditions — Ischemia; Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug Eluting Balloon (Experimental)
  Interventions: Device: drug eluting balloon

INTERVENTIONS:
Device: drug eluting balloon — drug eluting balloon bifurcated coronary lesions single arm study

SUMMARY:
The aim of the study is to investigate the feasibility of Paclitaxel-eluting PTCA-balloon dilation (SeQuent Please) followed by bare metal stent (Coroflex ) deployment in the main branch (reference diameter: ≥ 2.5 mm and ≤ 3.8 mm, reference diameter of side branch: ≥ 2.0 mm and ≤ 3.5 mm, length of stenoses in either branch ≤ 20 mm) in the treatment of significant (>70%) de-novo-bifurcation stenoses of any Medina classification type in the native left coronary artery as reflected by procedural success and to evaluate the preservation of vessel patency.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable angina pectoris (CCS class 1-3) or with unstable angina pectoris (Braunwald class 1-2, A-C) or documented ischemia or with documented silent ischemia
* Women of childbearing potential may not be pregnant nor have the desire to becoming pregnant during the first year following the study procedure. Hence, patients will be advised to use an adequate birth control method up to and including 6-month follow-up
* Patients who are mentally and linguistically able to understand the aim of the study and to show sufficient compliance in following the study protocol
* Patients must agree to undergo the 9-month angiographic follow-up
* Patients must agree to undergo the 3-year clinical follow-up
* Patient is able to verbally acknowledge and understand the associated risks, benefits, and treatment alternatives of this trial. The patients, by providing their informed consent, must agree to these risks and benefits as stated in the patient informed consent document.

Inclusion Criteria: Lesion Related

* De-novo bifurcational native left coronary artery lesion (reference diameter LAD or LCx: 2.5 mm to 3.8 mm, length of stenosis: ≤ 20 mm, reference diameter D1/D2 or OMS1/OMS2: 2.0 mm to 3.5 mm, length of stenosis: ≤ 20 mm)
* Diameter stenosis pre procedure must be either more then 70 % in either one or both branches of the lesion (i.e., bifurcational lesion of any type of the Medina classification) or more then 50 % if ischemia corresponding to the target lesion is documented either by exercise stress ECG, stress echocardiography, scintigraphy, MRT, or suspected based on angina pectoris
* Single or multi-vessel coronary artery disease

Exclusion Criteria:

* Patients with acute (< 24 h) or recent (48 hours) myocardial infarction
* Patients with unstable angina pectoris (Braunwald class 3)
* Patients with severe congestive heart failure
* Patients with severe heart failure NYHA IV
* Patients demonstrating clinical signs of cardiogenic shock at the time of the procedure (systolic blood pressure of less than 80 mmHg requiring inotropic support, IABP, and/or fluid challenge)
* Patients with severe valvular heart disease
* Women who are pregnant or lactating
* Patients with life expectancy of less than five years or factors making clinical follow-up difficult
* Patients with bleeding diathesis in whom anticoagulation or anti-platelet medication is contraindicated
* Patients who had a cerebral stroke < 6 months prior to the procedure
* Patient participates in other clinical trials involving any investigational device or drug
* Untreated hyperthyroidism
* Patient has presence or history of severe renal failure (GFR<30ml/min, "Cockcroft Gault") and is therefore at high risk for angiography associated renal complications. Patient's serum creatinine levels must be documented
* Post transplantation of any organ or immune suppressive medication
* Other disease to jeopardize follow-up (e.g., malignancy)
* Addiction to any drug or to alcohol
* Patients with any type of surgery during the week preceding the interventional procedure.
* Therapy with anticoagulants

Exclusion Criteria: Lesion Related

* Evidence of extensive thrombosis within target vessel before the intervention
* Multilesion percutaneous coronary intervention beside the bifurcation lesion in the left coronary artery (no other intervention is admitted during the same procedure)
* Patients with another coronary stent implanted previously into the target vessel ≤ 15 mm distant to the current lesion, drug eluting stents less than 9 months and bare metal stents or stents with passive coatings less than 3 months before the PEPCAD V BIF
* Target lesion located in any type of coronary bypass (i.e., venous graft, arterial bypass) or graft/native artery connection
* Coronary artery occlusion of any type (e.g., acute or chronic)
* In-stent restenosis
* In-segment restenosis of the native vessel within 4 mm adjacent to the target lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-10; Primary Completion 2011-05 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Procedural success (main branch ≤ 30%, side branch ≤ 50%, TIMI Flow 3) | acute

SECONDARY OUTCOMES:
In-segment late lumen loss at 9 months in either branch | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: D. G. Mathey, MD, Principal Investigator — Hamburg University Cardiovascular Center GmbH; F. X. Kleber, MD, Principal Investigator — Department of Internal Medicine Unfallkrankenhaus Berlin
Locations (2):
- Germany (2):
  - F.X.Kleber, Berlin
  - D.G: Mathey, Hamburg